CLINICAL TRIAL: NCT07343427
Title: Central Sensitization and Migraine Disability Following Greater Occipital Nerve Pulsed Radiofrequency: A Prospective Observational Study
Brief Title: Impact of GON PRF on Central Sensitization in Migraine Patients
Acronym: GON PRF-CS
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Ankara City Hospital Bilkent (Other)
Responsible Party: Principal Investigator, Gülçin Babaoğlu, Medical doctor, pain specialist, Ankara City Hospital Bilkent
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: TABED 2-25-979
Record Dates: First submitted 2026-01-07; First posted 2026-01-15 (Actual); Last update posted 2026-01-21 (Actual); Status verified 2026-01

CONDITIONS: Migraine; Central Sensitization
Keywords: Migraine; Central sensitization; Greater occipital nerve; Pulsed radiofrequency
MeSH Terms: conditions — Migraine Disorders

STUDY DESIGN:
Intervention Model Description: This is a single-group, prospective interventional study in which all enrolled participants undergo ultrasound-guided pulsed radiofrequency of the greater occipital nerve as part of routine clinical care. Clinical and patient-reported outcomes are assessed at baseline and at 1 and 3 months following the intervention to evaluate within-subject changes over time. No control or comparator group is included.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Greater Occipital Nerve Pulsed Radiofrequency (Experimental): Participants assigned to this arm will undergo ultrasound-guided pulsed radiofrequency of the greater occipital nerve as part of routine clinical care. The procedure will be performed under sterile operating room conditions with standardized pulsed radiofrequency parameters, maintaining electrode tip temperature at or below 42°C. Clinical and patient-reported outcomes will be assessed at baseline and at 1 and 3 months following the intervention.
  Interventions: Procedure: Greater occipital nerve radiofrequency

INTERVENTIONS:
Procedure: Greater occipital nerve radiofrequency — Ultrasound-guided pulsed radiofrequency will be applied to the greater occipital nerve under sterile operating room conditions. Participants will be positioned prone with the neck in flexion. Using a linear ultrasound transducer, the greater occipital nerve will be identified in the fascial plane between the obliquus capitis inferior and semispinalis capitis muscles at the C2 level. A 22-gauge radiofrequency cannula with a 5-mm active tip will be advanced using an in-plane technique toward the target nerve. Correct positioning will be confirmed by sensory stimulation at low voltage. Pulsed radiofrequency will be delivered at 45 V for 360 seconds with a pulse frequency of 5 Hz and pulse width of 5 ms, while maintaining the electrode tip temperature at or below 42°C. Participants will be monitored during and after the procedure according to standard clinical practice.

SUMMARY:
Background: Central sensitization and cutaneous allodynia are key mechanisms implicated in migraine chronification and disability. Pulsed radiofrequency (PRF) of the greater occipital nerve (GON) has emerged as a neuromodulatory intervention for refractory headache disorders; however, its effects on central sensitization remain insufficiently characterized.

Objective: To prospectively evaluate changes in central sensitization, allodynia, and migraine-related disability following GON pulsed radiofrequency in patients with migraine.

Methods: In this prospective observational study, adult patients with episodic or chronic migraine undergoing ultrasound-guided GON pulsed radiofrequency were evaluated at baseline and at 1 and 3 months post-procedure. Central sensitization was assessed using the Central Sensitization Inventory (CSI), cutaneous allodynia using the Allodynia Symptom Checklist (ASC-12), and migraine-related disability using the Migraine Disability Assessment Scale (MIDAS). Monthly headache days and acute medication use were also recorded.

Results: Changes in CSI, ASC-12, MIDAS scores, headache frequency, and acute medication use over follow-up were analyzed using repeated-measures statistical methods.

Conclusions: This study provides prospective data on sensory and clinical outcomes following GON pulsed radiofrequency, contributing to the understanding of its potential role in modulating central sensitization in migraine.

DETAILED DESCRIPTION:
Migraine is a highly prevalent neurological disorder associated with substantial disability, reduced quality of life, and significant socioeconomic burden. Increasing evidence indicates that migraine chronification is closely linked to central sensitization, characterized by enhanced excitability of central nociceptive pathways, impaired pain modulation, and the clinical manifestation of cutaneous allodynia. Persistent central sensitization is considered a key mechanism underlying increased attack frequency, treatment refractoriness, and migraine-related disability.

The greater occipital nerve (GON), originating from the dorsal ramus of the C2 spinal nerve, provides sensory innervation to the occipital region and has direct anatomical and functional connections with the trigeminocervical complex. Modulation of afferent input from the GON has been shown to influence trigeminal nociceptive processing, supporting its role as a therapeutic target in migraine and other primary headache disorders. Although GON blocks may reduce headache burden, their effects are typically transient, highlighting the need for longer-lasting neuromodulatory strategies.

Pulsed radiofrequency (PRF) is a minimally destructive neuromodulation technique that delivers short bursts of high-voltage electrical current while maintaining tissue temperatures below neurodestructive thresholds. Unlike continuous radiofrequency ablation, PRF is believed to exert its effects through neuromodulatory mechanisms rather than structural nerve injury. Previous studies have suggested that GON-targeted PRF may reduce headache frequency and intensity; however, data regarding its effects on central sensitization and sensory amplification in migraine remain limited.

This prospective observational study is designed to evaluate changes in central sensitization, cutaneous allodynia, and migraine-related disability following ultrasound-guided GON pulsed radiofrequency in patients with episodic or chronic migraine. Adult patients meeting International Classification of Headache Disorders, 3rd edition (ICHD-3) criteria for migraine and scheduled for GON PRF as part of routine clinical care will be enrolled. All procedures will be performed under sterile operating room conditions using ultrasound guidance to identify the GON between the obliquus capitis inferior and semispinalis capitis muscles. PRF will be applied with standardized parameters, maintaining electrode tip temperature at or below 42°C.

Participants will undergo clinical assessments at baseline and at 1 and 3 months after the procedure. Central sensitization will be assessed using the Central Sensitization Inventory (CSI), cutaneous allodynia using the Allodynia Symptom Checklist (ASC-12), and migraine-related disability using the Migraine Disability Assessment Scale (MIDAS). In addition, monthly moderate and severe headache days and acute migraine medication use will be recorded. Adverse events related to the procedure will be systematically monitored throughout the follow-up period.

By prospectively evaluating sensory and clinical outcomes over time, this study aims to provide detailed observational data on the potential neuromodulatory effects of GON pulsed radiofrequency on central sensitization and migraine-related disability. The findings are expected to contribute to a better understanding of patient-reported sensory changes following GON PRF and to inform future controlled studies investigating neuromodulation-based interventions in migraine.

ELIGIBILITY:
Inclusion Criteria:

* Adults aged 18 years or older

Diagnosis of episodic or chronic migraine according to the International Classification of Headache Disorders, 3rd edition (ICHD-3)

Planned to undergo ultrasound-guided greater occipital nerve pulsed radiofrequency as part of routine clinical care

Ability to complete self-reported questionnaires (CSI, ASC-12, MIDAS)

Willingness and ability to provide written informed consent

Exclusion Criteria:

* Presence of other primary headache disorders (e.g., cluster headache, tension-type headache as the primary diagnosis)

Secondary headache disorders, including headache attributed to structural, infectious, inflammatory, or vascular causes

Prior greater occipital nerve pulsed radiofrequency treatment within the past 12 months

History of cervical spine surgery, significant cervical trauma, or structural pathology that may interfere with the procedure

Known coagulopathy or current use of anticoagulant therapy that cannot be safely interrupted

Local infection at or near the planned injection site

Severe uncontrolled psychiatric or neurological disorders that may impair study participation or questionnaire reliability

Pregnancy or breastfeeding

Inability to comply with follow-up visits or study procedures

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2026-02-01 (Estimated); Primary Completion 2026-06-01 (Estimated); Study Completion 2026-09-01 (Estimated)

PRIMARY OUTCOMES:
Change in Central Sensitization Inventory (CSI) Total Score | Baseline to 3 months after greater occipital nerve pulsed radiofrequency
  Change in central sensitization symptoms assessed using the Central Sensitization Inventory (CSI), a validated 25-item self-reported questionnaire with scores ranging from 0 to 100, where higher scores indicate greater symptom severity.

SECONDARY OUTCOMES:
Change in Allodynia Symptom Checklist (ASC-12) Score | Baseline to 1 month and 3 months after the procedure
  The Allodynia Symptom Checklist-12 (ASC-12) is a patient-reported outcome measure assessing the presence and severity of cutaneous allodynia during migraine attacks. The total score ranges from 0 to 24, with higher scores indicating more severe allodynia symptoms. This outcome is defined as the change in ASC-12 total score from baseline to 1 month and 3 months of follow-up.
Change in Migraine Disability Assessment Scale (MIDAS) Score | Baseline to 1 month and 3 months after the procedure
  The Migraine Disability Assessment (MIDAS) questionnaire evaluates headache-related disability over the past 3 months by quantifying the impact of migraines on work, household, and social activities. The total MIDAS score ranges from 0 to 270, with higher scores indicating greater migraine-related disability. This outcome is defined as the change in MIDAS total score from baseline to 1 month and 3 months of follow-up.
Change in Acute Migraine Medication Use | Baseline to 1 month and 3 months after the procedure
  Change in the number of days per month requiring acute migraine medication.
Adverse Events | Up to 3 months after the procedure
  Frequency and type of procedure-related adverse events recorded throughout the follow-up period.

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Oliveira K, Dhondt N, Englesakis M, Goel A, Hoydonckx Y. Pulsed Radiofrequency Neuromodulation of the Greater Occipital Nerve for the Treatment of Headache Disorders in Adults: A Systematic Review. Can J Pain. 2024 May 15;8(1):2355571. doi: 10.1080/24740527.2024.2355571. eCollection 2024. PMID 38915302
- [Result] Suzuki K, Suzuki S, Shiina T, Kobayashi S, Hirata K. Central Sensitization in Migraine: A Narrative Review. J Pain Res. 2022 Sep 7;15:2673-2682. doi: 10.2147/JPR.S329280. eCollection 2022. PMID 36101891
- [Result] GBD 2021 Nervous System Disorders Collaborators. Global, regional, and national burden of disorders affecting the nervous system, 1990-2021: a systematic analysis for the Global Burden of Disease Study 2021. Lancet Neurol. 2024 Apr;23(4):344-381. doi: 10.1016/S1474-4422(24)00038-3. Epub 2024 Mar 14. PMID 38493795